CLINICAL TRIAL: NCT00288652
Title: [S,S]-Reboxetine Dose-Range Finding Trial: A 16-Week, Randomized, Double-Blind, Placebo And An Active Comparator Controlled, Multi-Center Trial Of [S,S]-Reboxetine In Patients With Postherpetic Neuralgia (PHN)
Brief Title: [S,S]-Reboxetine Dose-Range Finding Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6061026
Record Dates: First submitted 2006-02-07; First posted 2006-02-08 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain | interventions — O-methyl reboxetine

INTERVENTIONS:
Drug: [S,S]-Reboxetine

SUMMARY:
The purpose of this study is to determine the effectiveness of different doses of [S,S]-Reboxetine in the treatment of chronic pain following a shingles infection

ELIGIBILITY:
Inclusion Criteria:

* Patients must have pain present for more than 3 months after the healing of shingles skin rash
* Patients at screening must have a score >/=40 mm on the pain visual analogue scale

Exclusion Criteria:

* Patients with significant renal and hepatic impairment
* Patients with other severe pain, that may impair the self-assessment of the pain due to shingles
* Patients with clinically abnormal electrocardiogram

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280
Dates: Start 2006-03; Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
The numerical pain intensity rating scale is used to assess pain and a change from baseline in pain score for week 14 will be calculated

SECONDARY OUTCOMES:
- The mean endpoint (week 14) sleep interference score change from baseline - Analysis of the Medical Outcomes Study Sleep Scale - Analysis of the Patient Global Impression of Change - Analysis of the SF-36 Health Survey

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (79):
- United States (79):
  - Pfizer Investigational Site, Huntsville, Alabama
  - Pfizer Investigational Site, Chandler, Arizona
  - Pfizer Investigational Site, Mesa, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Sun City, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Hot Springs, Arkansas
  - Pfizer Investigational Site, Arcadia, California
  - Pfizer Investigational Site, Fullerton, California
  - Pfizer Investigational Site, Irvine, California
  - Pfizer Investigational Site, Laguna Hills, California
  - Pfizer Investigational Site, Loma Linda, California
  - Pfizer Investigational Site, Orange, California
  - Pfizer Investigational Site, Redondo Beach, California
  - Pfizer Investigational Site, Whittier, California
  - Pfizer Investigational Site, Boulder, Colorado
  - Pfizer Investigational Site, Bradenton, Florida
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Fort Myers, Florida
  - Pfizer Investigational Site, Holly Hill, Florida
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Kissimmee, Florida
  - Pfizer Investigational Site, Largo, Florida
  - Pfizer Investigational Site, Longwood, Florida
  - Pfizer Investigational Site, Melbourne, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Oviedo, Florida
  - Pfizer Investigational Site, Palm Beach Gardens, Florida
  - Pfizer Investigational Site, Plantation, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Oak Brook, Illinois
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Topeka, Kansas
  - Pfizer Investigational Site, Ruston, Louisiana
  - Pfizer Investigational Site, Towson, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Brockton, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Southaven, Mississippi
  - Pfizer Investigational Site, Independence, Missouri
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Nixa, Missouri
  - Pfizer Investigational Site, Sprinfield, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Billings, Montana
  - Pfizer Investigational Site, Clifton, New Jersey
  - Pfizer Investigational Site, Hackensack, New Jersey
  - Pfizer Investigational Site, Teaneck, New Jersey
  - Pfizer Investigational Site, Sante Fe, New Mexico
  - Pfizer Investigational Site, Albany, New York
  - Pfizer Investigational Site, Amherst, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Orchard Park, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Asheville, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Fargo, North Dakota
  - Pfizer Investigational Site, Canfield, Ohio
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Columbus, Ohio
  - Pfizer Investigational Site, Kettering, Ohio
  - Pfizer Investigational Site, Toledo, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Allentown, Pennsylvania
  - Pfizer Investigational Site, Altoona, Pennsylvania
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Jackson, Tennessee
  - Pfizer Investigational Site, Kingsport, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Norfolk, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Seattle, Washington
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Tacoma, Washington

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6061026&StudyName=%5BS%2CS%5D%2DReboxetine+Dose%2DRange+Finding+Trial